CLINICAL TRIAL: NCT01835639
Title: Pilot Study: Efficacy and Safety of Vitamin D Supplementation in Glomerular Disease
Brief Title: Vitamin D Supplementation in Glomerular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); American Society of Nephrology (Other); The NephCure Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-009753; K23DK093556 (NIH)
Record Dates: First submitted 2013-04-17; First posted 2013-04-19 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Glomerular Disease
Keywords: Glomerular Disease; Vitamin D; Steroid-resistant nephrotic syndrome; Minimal change disease; Focal segmental glomerulosclerosis (FSGS); Membranous Nephropathy; Membranoprolfierative Glomerulonephritis; immunoglobulin A (IgA) Nephropathy; FSGS; IgA Nephropathy
MeSH Terms: conditions — Nephrotic Syndrome; Nephrosis, Lipoid; Glomerulosclerosis, Focal Segmental; Glomerulonephritis, Membranous; Kidney Diseases; Glomerulonephritis, IGA | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vitamin D Supplementation (Experimental): Cholecalciferol, 2000 or 4000 IUs by mouth daily for 12 weeks
  Interventions: Dietary Supplement: Cholecalciferol, 2000 or 4000 IUs by mouth daily for 12 weeks

INTERVENTIONS:
Dietary Supplement: Cholecalciferol, 2000 or 4000 IUs by mouth daily for 12 weeks — Supplements will be provided as oral capsules.
  Other Names: Vitamin D

SUMMARY:
This multi-site, pilot study will assess vitamin D supplementation in children and young adults with Glomerular Disease. .

DETAILED DESCRIPTION:
Vitamin D deficiency has been linked to a variety of adverse health outcomes. Nephrotic patients have very low vitamin D levels, and the underlying mechanisms are not known. Furthermore, approaches to safely and effectively supplement vitamin D in these patients have not been established. The purpose of this research study is to learn if vitamin D supplementation is safe and effective in patients with primary glomerular disease and to also help establish the treatment guidelines. About 35 patients with primary glomerular disease, ages 5-30 years old, will take part in this study. Participants will be asked to take vitamin D supplements each day for 12 weeks and will have 3 study visits.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, age 5-30 years
* Diagnosis of primary glomerular disease (such as steroid-resistant nephrotic syndrome, minimal change disease, FSGS, membranous nephropathy, membranoprolfierative glomerulonephritis, and Immunoglobulin A [IgA] nephropathy) without systemic inflammatory disorders (i.e. lupus, vasculitis)
* Serum 25(OH)D level <30 ng/ml and urine protein:creatinine ratio ≥0.5 at Screening Visit.

Exclusion Criteria:

* Pregnancy
* estimated Glomerular Filtration Rate (eGFR) <30 ml/min/1.73m2 at Screening Visit
* Serum phosphorus > 5.5 mg/dl or hypercalcemia
* Chronic medical conditions or medications unrelated to the renal disease that may impact vitamin D status
* Known history of kidney stone(s)

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2013-04; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of vitamin D supplementation, by the increase in total and free 25(OH)D levels. | 12 weeks
To assess the safety of vitamin D supplementation, by serum Ionized calcium (ICal), Pi, and 25(OH)D, and urinary calcium excretion. | 12 weeks

SECONDARY OUTCOMES:
To assess the innate immune response, measured by changes in the induction of Human cathelicidin antimicrobial protein (hCAP) in human monocytes. | 12 weeks
To assess intra-renal inflammation, measured by changes in urinary Macrophage chemo-attractant protein 1 (MCP-1). | 12 weeks
To assess arterial stiffness, measured by changes in pulse wave velocity. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Denburg, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (5):
- United States (5):
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Johns Hopkins University,Division of Pediatric Nephrology, Baltimore, Maryland
  - North Shore-Long Island Jewish Health System, New Hyde Park, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania